CLINICAL TRIAL: NCT02477813
Title: Phase II Trial of Temozolomide in Patients Affected by Relapsed Sensitive or Refractory Small Cell Lung Cancer With MGMT Methylation (TeRes). GOPAV03
Brief Title: Temozolomide in Patients Affected by Relapsed Sensitive or Refractory Small Cell Lung Cancer With MGMT Methylation
Acronym: TeRes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of eligible patient recruitment
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST162.09
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Small Cell Lung Cancer Recurrent
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temozolomide (Experimental): oral Temozolomide 200 mg/m2/die for 5 consecutive days, every 28 days.Treatment will be continued until tumor progression, intolerable toxicity or patient refusal
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — 200 mg/m2 die for 5 consecutive days every 28 days. Treatment will be continued until tumor progression, intolerable toxicity or patient refusal

SUMMARY:
It is a single-arm, open label clinical trial. Patients affected by relapsed or refractory small-cell lung cancer patients with MGMT promoter methylation are included in this study; they will be treated with oral Temozolomide 200 mg/m2 die for 5 consecutive days every 28 days. Treatment will be continued until tumor progression, intolerable toxicity or patient refusal.

A Minimax Simon 2-stage design will be used. - First stage: 9 patients If 1 or less responses will be observed, the trial will be ended.- Second stage: other 10 patients (for a total of 19 subjects enrolled) If 5 or less responses will be observed in 19 patients, the treatment will not be considered active, while if 6 or more responses will be observed, the treatment will be considered sufficiently active to warrant further testing. Since the rate of methylation ranges from 20 to 48% the number of patients to be screened should be between 40 and 95.

The primary objective is to determine the overall response rate [ORR = CR + PR]; the secondary objectives are to determine the time to Progression (TTP), the overall Survival (OS), the toxicity and the correlation between response Rate (RR) and the level of MGMT promoter methylation and/or base excision repair (BER) genes alterations.

DETAILED DESCRIPTION:
This is a single-arm, open-label, phase II study. Patients must have histologically or cytologically confirmed small cell lung cancer (SCLC), both limited or extensive disease, relapsed after one or two prior chemotherapy regimens MGMT promoter methylation status will be evaluated on a histological tissue sample (after patient signature of a specific informed consent form for this biological evaluation) using Pyrosequencing technique and the main 10 CpG islands of MGMT promoter will be studied. Only patients with MGMT promoter methylation will be enrolled in the clinical trial. To be eligible patients may have received 1 or 2 prior chemotherapeutic regimens. Patients with brain metastases may be enrolled.

Patients will be informed about the palliative nature of the treatment . Patients will be treated with oral Temozolomide 200 mg/m2/die for 5 consecutive days .

Treatment will be repeated every 28 days and continued until disease progression, intolerable toxicity or patient refusal.

Response to chemotherapy will be monitored every three cycles by CT scan of the chest and the abdomen and computed tomography scan or magnetic resonance imaging of the whole brain. Response to treatment will be evaluated according to RECIST 1.1 criteria.

In case of progressive disease (PD) the patients will discontinue treatment. In case of stable disease (SD), partial response (PR) or complete response (CR) patients continue treatment until disease progression, intolerable toxicity or patient refusal.

After the end of treatment, if disease progression will not occur, patients will be evaluated every 3 months by CT scan of the chest and the abdomen and CT scan or RM of the whole brain until disease progression.

Planned follow-up visits will continue until disease progression and patients will be monitored for survival and toxicity .

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC with MGMT methylation.
* Patient previously treated by one or two chemotherapy lines.
* Age ≤ 75 and Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
* Patients must have measurable disease, defined as at least one lesion than can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20mm with conventional techniques or as >10mm with spiral CT scan.
* Patient with controlled brain metastases are eligible.
* Patient previously treated with chest and/or brain RT are eligible.
* Life expectancy >3 months.
* Patient must have normal organ and marrow function as defined below: leukocytes >3,000/μL, absolute neutrophil count >1,000/μL, platelets>100,000/μL, total bilirubin within normal institutional limits, AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal, creatinine within normal institutional limits
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the study and for 3 months thereafter.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Histologically or cytologically confirmed SCLC without MGMT methylation.
* Patients who have received three or more previous chemotherapy lines for small cell lung cancer or radiotherapy on target lesions.
* Symptomatic uncontrolled CNS metastasis.
* Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
* Presence of infection.
* History or evidence of malabsorption syndrome or disease that may significantly affect gastrointestinal function.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide or other agents used in the study.
* Presence of medical problems of sufficient severity to prevent full compliance with the study.
* Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR): | from randomization up to 3 years
  The percentage of patients whose cancer achieve either a partial response or a complete response

SECONDARY OUTCOMES:
Time to tumor progression (TTP) | from randomization up to 36 months
  It is defined as the time from registration until objective tumor progression NOT including death. Patients died for any cause or who are lost at follow up are censored.
Overall survival time (OS): | from randomization up to 36 months
  Time from enrolment to the date of death. For subjects with no known date of death, survival time will be censored at the date of their last on-study assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Casanova, MD, Principal Investigator — Oncology Department, PO Ravenna, AUSL della Romagna
Locations (8):
- Italy (8):
  - Ircc Irst, Meldola, FC
  - Oncologia Medica, Azienda ospedaliera universitaria di Ferrara, Ferrara, FE
  - Oncologia Medica AOU Policlinico di Modena, Modena, MO
  - U.O. Oncologia Medica, Faenza, RA
  - U.O Oncologia medica, Lugo, RA
  - UO Oncologia Medica, Ospedale S.Maria delle Croci, Ravenna, RA
  - U.O Oncologia medica, Rimini, RN
  - Oncologia Medica Ospedale Guglielmo da Saliceto, Piacenza